CLINICAL TRIAL: NCT00375700
Title: Efficacy of an Oral Nutrition Supplement on the Total Caloric and Protein Intake of Head and Neck Cancer Patients During the Last 2 Weeks of Radiation Therapy
Brief Title: Effect of an Oral Supplement on the Total Energy and Protein Intake of Head and Neck Cancer Patients in the Last 2 Weeks of Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN-4-0029 / 23027
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-03

CONDITIONS: Head and Neck Cancer
Keywords: food; diet; oral supplement; head and neck cancer; radiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement

SUMMARY:
In this study, an oral nutrition supplement has been developed that take into consideration: the nutritional requirements, treatment side-effects and taste preferences of head and neck cancer patients; the acceptance of a supplement when experiencing radiation therapy side-effects; and the taste preferences of head and neck cancer patients which may affect the supplement intake. We hope to increase dietary intake during the last 2 weeks of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosed with head and neck cancer including the lip, oral cavity, salivary glands, paranasal sinuses, oropharynx, nasopharynx, hypopharynx, larynx and thyroid.
* all histologic types of cancer
* all tumour stages according to American Joint Committee for Cancer (AJCC) Staging
* all forms of RT including standard or investigational for head and neck cancers
* alert and mentally competent
* English speaking

Exclusion Criteria:

* an allergy or intolerance to any of the substances used in the nutrition supplement
* Type I or II diabetes mellitus
* renal insufficiency
* unable to swallow
* additional criteria of all forms of chemotherapy standard or investigational or combination of radiation/chemotherapy standard or investigational for head and neck cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
total energy and protein intake | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Kubrak, PhD, Principal Investigator — University of Alberta